CLINICAL TRIAL: NCT03708146
Title: A Double-Blind, Randomised, Placebo-Controlled, Parallel Group Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of BIA 5 1058 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BIA 5-1058
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-51058-116; 2018-000113-20 (EudraCT Number)
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Disease+Pulmonary Disease; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Cohort 1 (BIA 5-1058 /50 mg/fasted) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 50 mg (as 2 x 25 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 2 (BIA 5-1058 /25 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 25 mg (as 1 x 25 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 3 (BIA 5-1058 /100 mg/fasted) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 100 mg (as 1 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 4 (BIA 5-1058 /50 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 50 mg (as 2 x 25 mg tablet) or matching placebo 12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 5 (BIA 5-1058 /150 mg/fasted) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 150 mg (as 1 x 100 mg and 2 x 25 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 6 (BIA 5-1058 /75 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 75 mg (as 3 x 25 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 7 (BIA 5-1058 /200 mg/fasted) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 200 mg (as 2 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 8 (BIA 5-1058 /100 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 100 mg (as 1 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 9 (BIA 5-1058 /400 mg/fasted) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 400 mg (as 4 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 10 (BIA 5-1058 /200 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 200 mg (as 2 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo
- Cohort 11 (BIA 5-1058 /400 mg/fed) (Experimental): 15 Subjects: 12 active and 3 placebo; BIA 5-1058 Tablet 400 mg (as 4 x 100 mg tablet) or matching placebo tablet (12 active and 3 placebo)
  Interventions: Drug: BIA 5-1058; Drug: Placebo

INTERVENTIONS:
Drug: BIA 5-1058 — 25 mg and 100 mg tablets; Oral, once-daily, from Day 1 to Day 10. In Cohorts 1, 3, 5, 7 and 9 (fasted), BIA 5-1058 will be orally administered in the morning after a minimum of 8 h fast. Subjects will remain fasted until 4 h post-dose and will receive lunch approximately 4 h after dosing.
  In Cohorts 2, 4, 6, 8 and 10 (fed), BIA 5-1058 will be orally administered in the morning after a moderate breakfast (containing approximately 550 kcal with fat contributing approximately 150 kcal). The meal should be consumed over a maximum period of 25 min, with dosing occurring 30 min after the start of the meal.
  Each dose will be administered with 240 mL water.
  Other Names: Zamicastat
Drug: Placebo — matching placebo tablet; Oral, once-daily, from Day 1 to Day 10. In Cohorts 1, 3, 5, 7 and 9 (fasted), placebo will be orally administered in the morning after a minimum of 8 h fast. Subjects will remain fasted until 4 h post-dose and will receive lunch approximately 4 h after dosing.
  In Cohorts 2, 4, 6, 8 and 10 (fed), placebo will be orally administered in the morning after a moderate breakfast (containing approximately 550 kcal with fat contributing approximately 150 kcal). The meal should be consumed over a maximum period of 25 min, with dosing occurring 30 min after the start of the meal.
  Each dose will be administered with 240 mL water.

SUMMARY:
This is a single centre, double-blind, randomised, placebo-controlled, parallel staggered group study of BIA 5-1058 in 11 different cohorts of 15 healthy subjects. Subjects will be randomly assigned to receive once-daily oral doses of BIA 5-1058 or matching placebo for 10 days.

The primary objectives of the study are to assess the safety and tolerability of BIA 5-1058 after repeated ascending doses under fed and fasted conditions and to assess the pharmacokinetics (PK) of BIA 5-1058 after repeated ascending doses under fed conditions having matching fasting cohorts for comparison of bioavailability.

It is planned that comparison cohorts will be dosed in parallel, i.e. Cohorts 1 and 2, 3 and 4, 5 and 6, 7 and 8 and 9 and 10. Cohorts may be split or dosed sequentially for logistical purposes; however, data from both comparison cohorts (e.g. Cohorts 1 and 2) must be available before dose escalation to the next dose levels.

DETAILED DESCRIPTION:
Each cohort will follow the same study design. Subjects will be screened for inclusion in the study between 28 and 3 days before the first dose. Eligible subjects will be admitted 2 days before dosing (Day -2) for all regimens, and will remain resident in the clinic until 72 h after the last dose (Day 13). On Day -1, blood samples will be taken in all cohorts for PD assessments at pre-defined time points. These time points will be time matched to Day 1 PK and PD time points. Subjects in Cohorts 2, 4, 6, 8, 10 and 11 (fed cohorts) will also undergo continuous cardiac monitoring via 24 h Holter recordings on Day -1.

Subjects in Cohorts 1, 3, 5, 7 and 9 will receive oral doses of BIA 5-1058 or matching placebo once daily from Day 1 to Day 10, administered in the morning of each day after a minimum of 8 h fast and will remain fasted until 4 h post-dose. Subjects in Cohorts 2, 4, 6, 8, 10 and 11 will receive oral doses of BIA 5-1058 or matching placebo once daily from Day 1 to Day 10, administered in the morning of each day, 30 minutes after the start of a moderate breakfast containing approximately 550 kcal with fat contributing approximately 150 kcal.

ELIGIBILITY:
Inclusion Criteria:

Able and willing to comply with the study restrictions and to give written informed consent before any study procedure; Male or non-pregnant, non-lactating female subjects aged 18 to 55 years, inclusive; Body mass index (BMI) between 18.0 and 32.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator; Healthy as determined by the investigator based on medical history, physical examination, clinical laboratory test results, vital signs (systolic blood pressure ≥ 90 mmHg and ≤ 150 mmHg, diastolic blood pressure ≥ 50 mmHg and ≤ 90 mmHg) and digital 12-lead ECG); Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibodies (HCV Ab) and anti-human immunodeficiency virus antibodies (HIV-1 and HIV-2 Ab) at screening; Clinical laboratory test results clinically acceptable at screening and admission Negative screen for alcohol and drugs of abuse at screening and admission Non-smokers or ex-smokers for at least 3 months;

Must adhere to the contraception requirements:

Male subjects and female partner willing to a condom plus an approved method of effective contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from the time of informed consent until 90 days after last dose of IMP. Male subjects must refrain from donating sperm throughout the study and for 90 days after the last dose of IMP; Female subjects of childbearing potential willing to use, with their partner, a condom and an approved method of highly effective contraception from the time of informed consent until 30 days after the last follow-up visit. Hormonal contraceptives are not permitted for female subjects. Female subjects must not donate ova from the time of the first dose until 90 days after the last dose of study drug; If female, nonchildbearing potential by reason of surgery or at least 1 year post menopause (i.e., 12 months post-last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing Negative serum pregnancy test at screening and negative urine pregnancy test on admission (all female subjects).

Exclusion Criteria:

Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders; Clinically relevant surgical history based on medical judgement by the investigator, excluding, for example, simple appendectomy or herniorrhaphy; Estimated glomerular filtration rate < 70 mL/min History of drug hypersensitivity or a presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active; Clinically relevant history of alcoholism or drug abuse in the past 5 years; Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, or a 25 mL of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type); Current smokers and those who have smoked within the last 3 months. A breath carbon monoxide reading of greater than 10 ppm at screening and admission; Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 3 months; Significant infection or known inflammatory process at screening or admission; Abnormal fundoscopy result at screening; Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission; Use of over the counter medications (including oral natural health products, vitamin and herbal supplements) in the 7 days before the first dose of IMP and use of prescription medications that may affect the safety or other study assessments, in the PI's opinion, are not permitted within 14 days before the first dose of IMP. By exception, acetaminophen/paracetamol ≤ 1 g/day is permitted. Other exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor; Subjects who have previously been enrolled in a BIA 5-1058 study or who have previously been enrolled and dosed in this study; Use of any investigational drug or participation in any clinical trial within 90 days prior to screening; Donation or reception of any blood or blood products within the 3 months prior to screening; Donation or loss of greater than 400 mL of blood within the previous 3 months; Vegetarians, vegans or other medical dietary restrictions; Subjects with a history of cholecystectomy or gall stones; Not able to communicate reliably with the investigator or sub-investigator; Unlikely to co-operate with the requirements of the study; Subjects who are study site employees, or immediate family members of a study site or sponsor employee; Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening; Females of childbearing potential who are pregnant or lactating (all female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test at admission); Males with pregnant partners; Failure to satisfy the investigator of fitness to participate for any other reason; Are unwilling or unable to give written informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Cmax: maximum observed concentration | Day 1, Day 6 and Day 10
  PK parameters analysis
Cmin: minimum observed concentration at steady state | Day 1, Day 6 and Day 10
  PK parameters analysis
Tlag: the elapsed time from dosing at which analyte was first quantifiable in a concentration vs time profile | Day 1, Day 6 and Day 10
  PK parameters analysis
Tmax: the time from dosing at which Cmax was apparent | Day 1, Day 6 and Day 10
  PK parameters analysis
AUC(0-t): area under the curve from 0 time to last measurable concentration | Day 1, Day 6 and Day 10
  PK parameters analysis
AUC(0-tau): area under the curve during a dosing interval | Day 1, Day 6 and Day 10
  PK parameters analysis
AUC(0-inf): area under the curve from 0 time extrapolated to infinity | Day 1, Day 6 and Day 10
  PK parameters analysis
AUC%extrap: percentage of AUC(0-inf) extrapolated beyond last measured time point | Day 1, Day 6 and Day 10
  PK parameters analysis
Lambda-z: the slope of the apparent elimination phase | Day 1, Day 6 and Day 10
  PK parameters analysis
t1/2: the apparent elimination half-life | Day 1, Day 6 and Day 10
  PK parameters analysis
Cl/F: clearance, the apparent volume cleared of parent drug per unit time after extravascular administration | Day 1, Day 6 and Day 10
  PK parameters analysis
MRT: mean residence time | Day 1, Day 6 and Day 10
  PK parameters analysis

SECONDARY OUTCOMES:
Emax: maximum observed % change from time-matched baseline | Day 1 and Day 10
  Pharmacodynamic parameters analysis
TEmax: Time of maximum observed % change from time-matched baseline | Day 1 and Day 10
  Pharmacodynamic parameters analysis
EAUC: % change from time-matched baseline area under the curve during a dosing interval | Day 1 and Day 10
  Pharmacodynamic parameters analysis
heart rate levels | pre-dose and Day 10
  Change from pre-submersion in heart rate levels following immersion of hand in ice cold water for 4 min (cold pressor test) - Cohort 9 only
Blood pressure levels | pre-dose and Day 10
  Change from pre-submersion in , blood pressure levels following immersion of hand in ice cold water for 4 min (cold pressor test) - Cohort 9 only
catecholamine (norepinephrine, epinephrine and dopamine) levels | pre-dose and Day 10
  Change from pre-submersion in , catecholamine (norepinephrine, epinephrine and dopamine) levels following immersion of hand in ice cold water for 4 min (cold pressor test) - Cohort 9 only
% inhibition of dopamine ß-hydroxylase (DβH) activity | Day 1 and Day 10

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided